CLINICAL TRIAL: NCT03215810
Title: A Phase I Clinical Trial Combining Nivolumab and Tumor Infiltrating Lymphocytes (TIL) for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Nivolumab and Tumor Infiltrating Lymphocytes (TIL) in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Prometheus Inc. (Industry); Stand Up To Cancer (Other); Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19122; CA209-9JA (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Non-Small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer; Squamous Cell Carcinoma; Advanced NSCLC; Adenosquamous Carcinoma; Adenocarcinomas
Keywords: Stage IV; NSCLC; Recurrent; TIL; Tumor-infiltrating Lymphocyte Therapy (TIL)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma, Adenosquamous; Adenocarcinoma; Recurrence | interventions — Nivolumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TIL+ Nivolumab (Experimental): Tumor-infiltrating Lymphocyte Therapy (TIL) + Nivolumab Treatment Plan: Tumor harvest, Tumor-infiltrating Lymphocytes growth, 4 cycles of nivolumab, cytoreductive chemotherapy with cyclophosphamide and fludarabine, TIL infusion, Interleukin-2 treatment.
  Interventions: Procedure: Tumor-infiltrating Lymphocytes (TIL); Drug: Nivolumab; Drug: Cyclophosphamide; Drug: Fludarabine; Other: Tumor-infiltrating Lymphocyte Therapy; Drug: Interleukin-2 (IL2)

INTERVENTIONS:
Procedure: Tumor-infiltrating Lymphocytes (TIL) — Tumor harvest for TIL growth in the lab: A sample of the participant's tumor will be collected and sent to the lab for TIL growth. TIL will be prepared and cryopreserved.
  Other Names: TIL
Drug: Nivolumab — Nivolumab will be administered intravenously at a fixed dose of 240 mg for 4 doses every 2 weeks prior to TIL. Nivolumab dose will be fixed at 480 mg every 4 weeks up to 12 months after TIL.
  Other Names: Opdivo
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 60 mg/kg/day IV in 250 mL normal saline (NS) over approximately 2 hours. Cyclophosphamide will be initiated seven days prior to the anticipated TIL transfer, and the precise timing will depend on the rate of in vitro TIL growth. The dose will be based on the patient's body weight, but to prevent undue toxicity, it will not exceed a dose greater than 140% of the maximum ideal body weight per Metropolitan Life Insurance Company, Height and Weight Table.
  Other Names: Cytoxan
Drug: Fludarabine — After administration of Cyclophosphamide, Fludarabine will then be infused at 25 mg/m^2 intravenous piggyback (IVPB) daily over approximately 30 minutes starting 5 days prior to TIL transfer. To prevent undue toxicity with fludarabine, the dose will be based on body surface area (BSA), but will not exceed a dose calculated on surface areas based on body weights greater than 140% of the maximum ideal body weight per Metropolitan Life Insurance Company Height and Weight Tables.
  Other Names: Fludara
Other: Tumor-infiltrating Lymphocyte Therapy — On day 0, all patients will receive TIL administered according to the current Moffitt Cell Therapy TIL Standard Operating Procedure (SOP). Eight (8) to twelve (12) hours after completing the TIL infusion, all participants will begin intermediate-dose decrescendo interleukin-2 (IL-2).
  Other Names: TIL
Drug: Interleukin-2 (IL2) — Interleukin-2 (IL-2) - a drug used to help the body's response to treatment on the immune system. A high dose regimen of IL-2 will be given after the infusion of the T-cells.
  Other Names: IL2; Proleukin®

SUMMARY:
Investigators plan to study the safety, side effects, and benefits of tumor-infiltrating lymphocytes (TILs) when they are given with the drug nivolumab. Nivolumab is a type of immunotherapy - a drug that is used to boost the ability of the immune system to fight cancer, infection, and other diseases.

DETAILED DESCRIPTION:
In this study, these special immune T-cells will be taken from a sample of the participant's tumor tissue that will be surgically removed. Certain parts of these cells will be multiplied, or grown, in the laboratory, using the drug interleukin-2 (IL-2) during part of the process. They will then be given back to the participant by an infusion in their veins. These cells are called tumor- infiltrating lymphocytes (TILs). The use of TILs involves a combination of drugs, including the following:

* Fludarabine and cyclophosphamide - two types of chemotherapy drugs. These drugs will be used for what is called lymphodepletion. The purpose of lymphodepletion in this study is to temporarily reduce the number of normal lymphocytes circulating in the participant's body before they are given the TILs that were grown in the lab. This is so that there will be more "space" for the lymphocytes (TILs) that will be infused in their veins.
* Interleukin-2 (IL-2) - a drug used to help the body's response to treatment on the immune system. A high dose regimen of IL-2 will be given after the participant receives the infusion of the T-cells.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to understand and give written informed consent
* Confirmed or suspected diagnosis of stage IV or recurrent non-small cell lung cancer (NSCLC). For suspected NSCLC, diagnosis must be histologically or cytologically confirmed prior to start of nivolumab treatment. Neuroendocrine cancers, or mixed neuroendocrine features in >10% of tumor cells, are excluded.
* Tumor deemed accessible by metastasectomy (TIL harvest) which expects to yield >1.5 cm^3 of resectable tumor amount.
* Measurable disease, even after resection of applicable lesion for TIL harvest. Defined as ≥1 lesion that is ≥10 mm in one dimension by CT scan, MRI, or calipers on clinical exam.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected survival > 6 months
* Patients with activating Epidermal Growth Factor Receptor (EGFR) mutation or Anaplastic Lymphoma Kinase (ALK) rearrangement which is expected to be responsive to available tyrosine kinase inhibitor therapy, must have been previously treated with an applicable tyrosine kinase inhibitor.
* Adequate normal organ and marrow function in an assessment performed within 7 days (+ 3 day window) of enrollment, defined as: Hemoglobin ≥ 9.0 g/dL; Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L (> 1000 per mm^3); Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3); Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) ≤ 1.5x the institutional upper limit of normal (ULN), (This will not apply to patients with confirmed Factor XII deficiency.); Serum bilirubin ≤ 1.5x the institutional ULN, or ≤ 3x ULN if confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology); Aspartate Aminotransferase (AST) (SGOT)/Alanine Aminotransferase (ALT) (SGPT) ≤ 2.5x institutional ULN unless liver metastases are present, in which case it must be ≤ 5x ULN; Serum creatinine of ≤ 1.5x institutional ULN; Albumin ≥ 2.5 g/dl.
* Positive screening Epstein Barr Virus (EBV) antibody titer on screening test.
* Cardiac stress test within past 6 months without evidence of reversible ischemia.
* Cardiac echocardiogram, stress test, or Multigated Acquisition Scan (MUGA) within past 6 months with demonstrated left ventricular ejection fraction (LVEF) > 50%
* Pulmonary function tests within past 6 months showing Diffusion Lung Capacity for Carbon Monoxide (DLCO) >50% of predicted. Adjusted DLCO based on hemoglobin concentration should be used, if available.

Exclusion Criteria:

* More than 5 lines of prior systemic therapy in the preceding 3 years.
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including but not limited to: nivolumab, atezolizumab, pembrolizumab, or durvalumab.
* Current or prior use of any immunosuppressive medications, such as corticosteroids, within 14 days before enrollment. a.) Oral hydrocortisone, only for the purposes of a documented and confirmed adrenal insufficiency diagnosis, is permitted if ≤ 25 mg daily total dose. b.) Inhaled, intranasal, or topical corticosteroids are permitted.
* Patients with untreated brain metastases. Treated brain metastases with radiation or surgery are allowed if: ≤ 3 cm in size AND ≤ 4 in number AND there is no evidence of progressive disease, on brain imaging ≥ 28 days after last day of central nervous system (CNS) treatment.
* History of leptomeningeal metastases.
* Current or prior use of anticancer therapy before TIL collection: a.) Chemotherapy within the past 4 weeks; b.) Tyrosine kinase inhibitor (TKI) within the past 1 week; c.) Investigational therapy within the past 4 weeks or 4 half-lives, whichever is shorter.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than stable atrial fibrillation) and significant carotid artery stenosis.
* Known to be HIV positive, hepatitis B or C positive, or both Rapid Plasma Reagin (RPR) and Fluorescent Treponemal Antibody (FTA positive). (Hepatitis B surface or core antibody alone is not indicative of Hepatitis B Virus (HBV) infection).
* Patients with rapidly progressing tumors, as judged by the investigator.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from electrocardiograms (ECGs) using Bazett's Correction
* Known history of previous tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to first anticipated dose of nivolumab.
* History of allogeneic organ transplant
* History of primary immunodeficiency
* History of severe hypersensitivity to nivolumab, cyclophosphamide, fludarabine, interleukin-2, or any excipient
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Patients with active systemic infections requiring intravenous antibiotics within 1 week prior to enrollment.
* Any unresolved toxicity (>CTCAE v4 grade 2) from previous anti-cancer therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy).
* History of pneumonitis or drug-related inflammatory lung disease
* Have a significant history of pulmonary disease that necessitates the use of supplemental oxygen, and patients with resting pulse oximetry less than 92% on room air.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, limited site eczema, or limited site plaque psoriasis not requiring systemic treatment (within the past 2 years), or other autoimmune conditions which are not expected to recur, are allowed after approval from the medical monitor or Principal Investigator (PI).
* Patients with other prior malignancies must have had a ≥ 2-year disease-free interval, except for: in situ carcinoma of the cervix, in situ ductal carcinoma of the breast, in situ prostate cancer, in situ bladder cancer. These must have been deemed stable and not expected to relapse. In addition, early stage skin cancers, including basal, squamous cell cutaneous carcinoma, and melanoma, are permitted if previously treated with curative intent and not expected to relapse.
* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until 4 months after conclusion of the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Creelan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - University of Florida Health Cancer Center., Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

REFERENCES:
- [Derived] Creelan BC, Wang C, Teer JK, Toloza EM, Yao J, Kim S, Landin AM, Mullinax JE, Saller JJ, Saltos AN, Noyes DR, Montoya LB, Curry W, Pilon-Thomas SA, Chiappori AA, Tanvetyanon T, Kaye FJ, Thompson ZJ, Yoder SJ, Fang B, Koomen JM, Sarnaik AA, Chen DT, Conejo-Garcia JR, Haura EB, Antonia SJ. Tumor-infiltrating lymphocyte treatment for anti-PD-1-resistant metastatic lung cancer: a phase 1 trial. Nat Med. 2021 Aug;27(8):1410-1418. doi: 10.1038/s41591-021-01462-y. Epub 2021 Aug 12. PMID 34385708

RESULTS

PARTICIPANT FLOW:
Groups:
- TIL+ Nivolumab: Nivolumab, 240 mg, IV infusion every 2 weeks for 8 weeks prior to Tumor Infiltrating Lymphocytes (TIL) infusion, and then after TIL infusion 480 mg every 4 weeks for up to 12 months
Period: Overall Study
Arm/Group | TIL+ Nivolumab
Started | 20
Completed | 16
Not Completed | 4
Not completed — Still responding to nivolumab | 1
Not completed — Insufficient TIL growth | 1
Not completed — Decline in performance status | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TIL+ Nivolumab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicity (DLT)
Description: Investigators plan to demonstrate that treatment with nivolumab in patients undergoing TIL therapy is safe with a continuous Pocock-type stopping boundary for serious toxicity of < 17%, with safety reported based upon Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria. DLT defined as: any grade ≥3 immune-related adverse event definitely attributable to nivolumab. DLT related to adoptive cell therapy will be defined as a non-hematologic grade 4 or higher adverse event that is immediately life-threatening occurring upon or after the start of therapy that is immediately life-threatening and not related to non-small cell lung cancer or other pre-existing condition. Safety: Toxicity will be assessed within 4 weeks of the adoptive TIL transfer. The accrual will be halted if excessive numbers of participants with toxicity are seen. For example, if there are 5 or more out of 10 participants (full follow-up) with toxicity, the trial will be stopped.
Time Frame: Up to 40 months
Population: All participants evaluable for safety
Measure: Number; unit: % participants w severe toxicity
Arm/Group | TIL+ Nivolumab
Number analyzed (Participants) | 16
% participants w severe toxicity | 17

2. Secondary Outcome: Number of Participants With Objective Response
Description: Participants displaying objective response associated with the treatment regimen per Response Evaluation Criteria in Solid Tumors (RECIST v.1.1). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: Up to 40 months
Population: Participants evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | TIL+ Nivolumab
Number analyzed (Participants) | 13
Participants
  Confirmed | 3
  Unconfirmed | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 years and 11 months
Description: Adverse Events includes all enrolled patients who started initial nivolumab (20) but only 16 received TIL. Therefore the denominator (20) includes all enrolled patients exposed to any study tx. This table is intended to represent a summary-level overview for all patients enrolled on the trial, and not intended to indicate attribution, frequency, or causality for specific drugs or TIL. Please refer to the publication for dedicated adverse event tables, including grade
Arm/Group | TIL+ Nivolumab
All-Cause Mortality (participants affected / at risk) | 7/20
Serious Adverse Events (participants affected / at risk) | 15/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIL+ Nivolumab (N=20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Systemic edema
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Fever (General disorders) | 3 (3)
Platelet count decreased (Investigations) | 2 (3)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1) — C-diff
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) — altered mental status related to polypharmacy
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Infections and infestations -Other (Infections and infestations) | 1 (1) — Thrush
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIL+ Nivolumab (N=20)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 10 (23)
Alkaline phosphatase increased (Investigations) | 14 (34)
Anemia (Blood and lymphatic system disorders) | 17 (151)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 11 (23)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (3)
Blood bilirubin increased (Investigations) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 2 (2)
Chills (General disorders) | 8 (13)
Cholesterol high (Investigations) | 1 (1)
Confusion (Psychiatric disorders) | 3 (4)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Creatinine increased (Investigations) | 6 (9)
Cytokine release syndrome (Immune system disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Delirium (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 16 (30)
Dizziness (Nervous system disorders) | 5 (6)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (21)
Edema cerebral (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 9 (9)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (2)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 12 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 10 (31)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (10)
Hematuria (Renal and urinary disorders) | 5 (8)
Hemoglobin increased (Investigations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (47)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 13 (40)
Hypermagnesemia (Metabolism and nutrition disorders) | 10 (19)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (64)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (54)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 13 (52)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (41)
Hypotension (Vascular disorders) | 10 (17)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Infections and infestations - Other (Infections and infestations) | 3 (3)
Infusion related reaction (General disorders) | 1 (1)
INR increased (Investigations) | 9 (20)
Insomnia (Psychiatric disorders) | 6 (8)
Investigations - Other (Investigations) | 5 (18)
Irregular menstruation (Reproductive system and breast disorders) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 18 (132)
Lymphocyte count increased (Investigations) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 15 (28)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (50)
Non-cardiac chest pain (General disorders) | 4 (4)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 10 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 15 (111)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (11)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Rhinitis infective (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 11 (18)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (4)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (3)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Vaginal infection (Infections and infestations) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (10)
Weight loss (Investigations) | 4 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4)
White blood cell decreased (Investigations) | 18 (97)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03215810/Prot_SAP_000.pdf